CLINICAL TRIAL: NCT05155111
Title: Telemedicine for Identification of Neonatal Encephalopathy
Brief Title: Telemedicine to Reduce Disparities in the Identification and Treatment of Neonatal Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Alexa Craig, Attending Neonatal and Pediatric Neurologist, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1781443
Record Dates: First submitted 2021-11-16; First posted 2021-12-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Neonatal Encephalopathy
Keywords: Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine arm (Experimental): Neonates will have telemedicine consultation to evaluate symptoms of neonatal encephalopathy
  Interventions: Diagnostic Test: Telemedicine consult

INTERVENTIONS:
Diagnostic Test: Telemedicine consult — A joint assessment between Neonatologist at bedside and Neurologist by telemedicine will be performed to assess severity of neonatal encephalopathy

SUMMARY:
This is a clinical trial using telemedicine as an intervention twice in the first 6 hours of life to assess neonatal encephalopathy, one of the key factors involved in the decision to treat a neonate with therapeutic hypothermia (TH). The investigators aim to enroll up to 30 neonates, anticipating that there will be about 5 neonates, who do not demonstrate moderate to severe neonatal encephalopathy, and therefore do not meet criteria for treatment with TH. The investigators will prospectively follow the clinical course of all 30neonates through monitoring with electroencephalogram (EEG) for up to 24 hours after birth to determine if seizures are present and by MRI of the brain prior to hospital discharge to determine if there is evidence of brain injury. Neonates will be enrolled in the study for the duration of their hospital admission.

DETAILED DESCRIPTION:
Neonatal encephalopathy is a clinically defined condition of disturbed neurological function in an infant of greater than 35 weeks gestation. Neonatal encephalopathy is most likely to occur following a traumatic birth that requires some degree of neonatal resuscitation. Therapeutic hypothermia (TH) is the standard-of-care neuroprotective therapy employed for neonates who have symptoms of moderate to severe neonatal encephalopathy. Assessment of neonatal encephalopathy can be challenging because the symptoms can fluctuate and because there is time pressure to decide to initiate TH before the neonate is 6 hours old, after which TH has almost no beneficial effect. Doctors struggle with the decision to treat neonates with milder symptoms and these neonates are at risk for two possible adverse outcomes; 1) an eligible neonate is not recognized and therefore not treated with TH or 2) an ineligible neonate may receive unnecessary treatment. The first error is one that can result in lifelong impairments such as learning delays, epilepsy and cerebral palsy for the untreated child and the second error, of unnecessary treatment is costly, invasive and not without risk of associated issues with morphine exposure, cold-induced injury to the skin or complications from venous access such as infection or blood clot.

In Maine, the investigators have successfully implemented telemedicine both in the tertiary care center and in the rural community hospital to permit visual evaluation of neonates and inform joint decision making in these challenging instances. Telemedicine provides the opportunity to have synchronous, unscheduled immediate expert consultation for neonatologists with pediatric neurology in the tertiary care center and for primary care physicians with both specialists in the community hospital setting. The objective of the present study is to develop the telemedicine consultative network to continue to improve patient selection for TH. The investigators aim to use telemedicine consults in three tertiary care centers (Maine Medical Center, Northern Light Eastern Maine Medical Center and the University of Vermont Medical Center) to develop evidence for the threshold at which neonates can be safely excluded from TH treatment. In Aim 1, the investigators will assess neonates with milder symptoms at least twice in the first 6 hours of life and for those not meeting criteria for moderate or severe neonatal encephalopathy, perform electroencephalogram (EEG) to rule out seizures and MRI of the brain to rule out injury. In aim 2, the investigators will compare the interrater reliability between the neonatologist neonatal encephalopathy exam and the one performed via telemedicine by the pediatric neurologist.

ELIGIBILITY:
Inclusion Criteria:

* Umbilical cord pH ≤7.0 or base deficit ≥ -16
* Umbilical cord pH 7.01 to 7.15 or base deficit between -10 and -16 AND one of the following;

  * a perinatal event, defined as severe fetal heart rate abnormality such as category 2 or 3 tracing with recurrent variable decelerations, prolonged decelerations or recurrent late decelerations, umbilical cord prolapse/rupture, uterine rupture, significant placental abruption, maternal trauma or hemorrhage or cardiopulmonary arrest)
  * 10-minute Apgar score < 5
  * Need for respiratory support for >10 minutes not otherwise due to a primary pulmonary process

Exclusion Criteria:

* Older than 6 hours
* Gestational age less than or equal to 35 6/7 weeks
* Birthweight <1800 grams
* Non-English speaking parents due to time constraints to perform the consent process

Ages: 0 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Combined outcome of seizure or brain Injury on imaging | First 10 days of life
  The primary outcome is a combined outcome. This will include the presence of absence of seizure activity on the electroencephalogram (EEG) during the first 24 hours of life and/or the presence or absence of injury to the brain detected on magnetic resonance imaging of the brain (MRI) performed prior to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Alexa K Craig, MD, Principal Investigator — physician
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No